CLINICAL TRIAL: NCT05357391
Title: Clinical Study of Pressure Injury Wound Prediction Model Using a Mobile Application System for Caring and Managing
Brief Title: Pressure Injury Prediction and Education Model Using a Mobile Application System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 110-113-E
Record Dates: First submitted 2022-01-05; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Pressure Injury; Wound
Keywords: Pressure injury; Wound prediction model; Mobile application system; Knowledge of wound care; Self-efficacy; Anxiety; Depression
MeSH Terms: conditions — Pressure Ulcer; Wounds and Injuries; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: 1. pressure injury prediction and education model group
  2. control group
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The pressure injury prediction and education model group (Experimental): The experimental group will be provided a pressure injury prediction of the patient and personalized care information of pressure injury by a smart care platform. The participants (primary caregivers) will fill out the questionnaires online at admission (baseline-T0) and before the patient is discharged(T1). The questionnaires will collect the following data, including demographic information(only T0), knowledge, self-efficacy, anxiety, depression of wound care(T0&T1), and satisfaction of the smart care platform(only T1). The time to fill out the questionnaires will be about 10 minutes.
  Interventions: Device: The Pressure Injury Prediction and Education model using a mobile application system
- The control group (No Intervention): Routine care

INTERVENTIONS:
Device: The Pressure Injury Prediction and Education model using a mobile application system — Data from the medical records will be used to analyze the probability and risk of wound healing for creating a Pressure Injury Prediction and Education Model using a mobile application system.
  Arms: The pressure injury prediction and education model group

SUMMARY:
Pressure injuries are common in the elderly and patients who reduced physical activities. Its complications significantly impact the health care system and social burden, even causing the death rate to be as high as 68%. This study aims to collect medical data regarding pressure injuries during hospitalization for developing the Pressure Injury Prediction and Education Model using a mobile application system. It can offer a prediction on the risk of pressure injury and be used as a teaching aid for pressure injury care, providing a personalized and evidence-based nursing information platform for patients, caregivers, and health professionals.

DETAILED DESCRIPTION:
This study will conduct a randomized controlled trial among 160 primary caregivers of patients with pressure injuries. They will be randomly assigned to the control group or the experimental group. In the control group, patients are routinely cared for in the ward, and this group will have no intervention. Routine care includes face-to-face training and educational pamphlets by the ward nurse. The experimental group will be provided a pressure injury prediction of the patient and personalized care information of pressure injury by a smart care platform. The participants (primary caregivers) will fill out the questionnaires online at admission (baseline-T0)and before the patient is discharged(T1). The questionnaires will collect the following data, including demographic information(only T0), knowledge, self-efficacy, anxiety, depression of pressure injury care(T0&T1), and satisfaction of the smart care platform(only T1). The time to fill out the questionnaires will be about 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. The primary caregiver for patients with pressure injury in the hospital.
2. The primary caregiver must be at least 20 years old, have clear consciousness, express independently, communicate in Mandarin and Taiwanese, use an Android phone by himself, and use a mobile phone application after explanation.

Exclusion Criteria:

The primary caregiver has a mental or cognitive impairment, cannot express consciousness clearly, or cannot operate mobile apps.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from the baseline score of the knowledge of pressure injury care to before discharge | Data will be collected on admission(baseline-T0) and before discharge(T1).
  The investigators designed the ten questions regarding pressure injury care knowledge to detect caregivers' understanding of pressure injury care. The higher scores reflect a greater understanding of pressure injury care.
Change from the baseline score of the pressure injury care self-efficacy of caregivers to before discharge | Data will be collected on admission(baseline-T0) and before discharge(T1).
  The fourteen items of the self-efficacy of pressure injury care are designed to detect caregivers' self-efficacy on pressure injury care. Response options on the items range from "no confidence" (1 point) to "every confidence" (5 points). The higher scores reflect greater self-efficacy on pressure injury care.
Change from the baseline score of the General Anxiety Disorder-7(GAD-7) to before discharge | Data will be collected on admission(baseline-T0) and before discharge(T1).
  The GAD-7 (Spitzer et al., 2006) is a one-dimensional instrument designed to detect generalized anxiety disorder symptoms defined in the DSM-IV. The item scores range from 0 (not at all) to 3 (nearly every day), resulting in a sum score ranging from 0 to 21. The higher scores reflect greater anxiety severity.
Change from the baseline score of the Patient Health Questionnaire-9(PHQ-9) to before discharge | Data will be collected on admission(baseline-T0) and before discharge(T1).
  The nine items of the PHQ-9 are designed to capture the nine Diagnostic and Statistical Manual of Mental Disorders (DSM) symptom criteria for a major depressive episode. Response options on the items range from "not at all" (0 points) to "nearly every day" (3 points). As a severity measure, the PHQ-9 score can range from 0 to 27.

SECONDARY OUTCOMES:
the satisfaction score of the smart care platform regarding pressure injury care | Data will be collected before discharge(T1).
  The ten items of satisfaction with the smart care platform are designed to detect caregivers' satisfaction with this platform. Response options on the items range from "strongly disagree " (1 point) to "strongly agree" (5 points), resulting in a sum score ranging from 10 to 50.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Ling Wu, BS, Principal Investigator — National Taiwan University Hospital Hsin-Chu Branch
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmad Zubaidi ZS, Ariffin F, Oun CTC, Katiman D. Caregiver burden among informal caregivers in the largest specialized palliative care unit in Malaysia: a cross sectional study. BMC Palliat Care. 2020 Dec 8;19(1):186. doi: 10.1186/s12904-020-00691-1. PMID 33292214
- [Background] Govina O, Vlachou E, Kalemikerakis I, Papageorgiou D, Kavga A, Konstantinidis T. Factors Associated with Anxiety and Depression among Family Caregivers of Patients Undergoing Palliative Radiotherapy. Asia Pac J Oncol Nurs. 2019 Jul-Sep;6(3):283-291. doi: 10.4103/apjon.apjon_74_18. PMID 31259225
- [Background] Santos CT, Almeida Mde A, Lucena Ade F. The Nursing Diagnosis of risk for pressure ulcer: content validation. Rev Lat Am Enfermagem. 2016 Jun 14;24:e2693. doi: 10.1590/1518-8345.0782.2693. PMID 27305182
- [Background] Wang Y, Chen R, Ding J, Yang L, Chen J, Huang B. Predictive value of pressure ulcer risk for obstructive coronary artery disease. Nurs Open. 2021 Jul;8(4):1848-1855. doi: 10.1002/nop2.835. Epub 2021 Mar 6. PMID 33675186
- [Background] Fishbein JN, Nisotel LE, MacDonald JJ, Amoyal Pensak N, Jacobs JM, Flanagan C, Jethwani K, Greer JA. Mobile Application to Promote Adherence to Oral Chemotherapy and Symptom Management: A Protocol for Design and Development. JMIR Res Protoc. 2017 Apr 20;6(4):e62. doi: 10.2196/resprot.6198. PMID 28428158
- [Background] Drew DA, Nguyen LH, Steves CJ, Menni C, Freydin M, Varsavsky T, Sudre CH, Cardoso MJ, Ourselin S, Wolf J, Spector TD, Chan AT; COPE Consortium. Rapid implementation of mobile technology for real-time epidemiology of COVID-19. Science. 2020 Jun 19;368(6497):1362-1367. doi: 10.1126/science.abc0473. Epub 2020 May 5. PMID 32371477